CLINICAL TRIAL: NCT00959569
Title: Esmolol in Cardiac Surgery. A Randomized Controlled Trial With Clinical
Brief Title: Esmolol in Cardiac Surgery
Acronym: BREVI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GO/URC/ER/mm 459/DG
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Surgery
Keywords: esmolol; cardiac surgery; cardiac anesthesia; mortality; beta blockers; beta-blockers; cardiac protection
MeSH Terms: interventions — esmolol; Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- esmolol (Experimental): the study group will receive esmolol (1-3 mg/kg)
  Interventions: Drug: Esmolol
- normosaline (Placebo Comparator): normosaline (same ml of the study drug)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esmolol — esmolol (1-3 mg/kg) during cardiac surgery
  Other Names: Beta-blocker; Beta blocker; breviblock
  Arms: esmolol
Drug: Placebo — normosaline (same ml of the study drug)
  Arms: normosaline

SUMMARY:
This large randomized double-blind clinical trial (esmolol vs placebo) will enroll patients undergoing cardiac surgery to study the additive cardiac protection of this therapeutic strategy.

ELIGIBILITY:
Inclusion Criteria:

* end diastolic diameter >60 mm and/or an ejection fraction <50%
* written informed consent
* age >18 years

Exclusion Criteria:

* previous unusual response to esmolol
* inclusion in other randomized studies
* esmolol administration in the previous 30 days
* emergency operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-08; Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of number of dead patients and/or number of patients requiring prolonged ICU stay. | Hospital stay (approximately 2 weeks)

SECONDARY OUTCOMES:
Number of patients with ventricular fibrillation after cardiopulmonary bypass | 30 days and 1 year
Number of patients with low cardiac output syndrome | 30 days and 1 year
Number of patients requiring post-operative inotropic support | 30 days and 1 year
peak postoperative cardiac troponin level | 30 days and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Vita-Salute University, Milan, Italy

REFERENCES:
- [Background] Zangrillo A, Turi S, Crescenzi G, Oriani A, Distaso F, Monaco F, Bignami E, Landoni G. Esmolol reduces perioperative ischemia in cardiac surgery: a meta-analysis of randomized controlled studies. J Cardiothorac Vasc Anesth. 2009 Oct;23(5):625-32. doi: 10.1053/j.jvca.2009.01.003. Epub 2009 Mar 18. PMID 19297196
- [Background] Crescenzi G, Rosica C, Marino G, Serini SM, Covello RD, Landoni G, Zangrillo A. The use of esmolol to treat systolic anterior motion of the mitral valve after mitral valve repair. Eur J Anaesthesiol. 2008 Apr;25(4):342-3. doi: 10.1017/S0265021507002876. No abstract available. PMID 18334040
- [Background] Landoni G, Zambon M, Zangrillo A. Reducing perioperative myocardial infarction with anesthetic drugs and techniques. Curr Drug Targets. 2009 Sep;10(9):858-62. doi: 10.2174/138945009789108837. Epub 2009 Sep 1. PMID 19538174
- [Background] Crescenzi G, Landoni G, Zangrillo A, Guarracino F, Rosica C, La Canna G, Alfieri O. Management and decision-making strategy for systolic anterior motion after mitral valve repair. J Thorac Cardiovasc Surg. 2009 Feb;137(2):320-5. doi: 10.1016/j.jtcvs.2008.08.018. PMID 19185145